CLINICAL TRIAL: NCT03062683
Title: Serum Lactate in Convulsive Syncopes Compared to Non-convulsive Syncopes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: Laktat-2017
Record Dates: First submitted 2017-02-20; First posted 2017-02-23 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-02

CONDITIONS: Syncope; Lactate Blood Increase
Keywords: lactate; syncope
MeSH Terms: conditions — Syncope; Hyperlactatemia | interventions — Lactic Acid; Prolactin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — repeated blood samples (2-5 ml)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-convulsive syncope patients: Patients with a non-convulsive syncope triggered by a tilting table examination and whose serum lactate, prolactin and creatine kinase conc. in blood samples had been measured after the event.
  Interventions: Other: Lactate, prolactin and creatine kinase conc.
- Convulsive syncope patients: Patients with a convulsive syncope triggered by a tilting table examination and whose serum lactate, prolactin and creatine kinase conc. in blood samples had been measured after the event.
  Interventions: Other: Lactate, prolactin and creatine kinase conc.

INTERVENTIONS:
Other: Lactate, prolactin and creatine kinase conc. — Lactate, prolactin and creatine kinase conc. in blood samples were measured

SUMMARY:
The investigators compared the serum lactate, serum prolactin and serum creatine kinase concentrations following convulsive and non-convulsive syncopes. The aim of the study was to investigate their importance as diagnostic markers in transient loss of consciousness.

DETAILED DESCRIPTION:
Unclear transient loss of consciousness is a frequent interdisciplinary diagnostic problem. Of particular importance is the distinction between epileptic and non-epileptic events. Our group showed in two previous studies that serum lactate is elevated in epileptic seizures, but mostly not in syncopes, psychogenic non-epileptic seizures and complex partial seizures. These results showed that lactate can be used as a diagnostic marker for the presence of a generalized epileptic seizure.It remains unclear whether a normal serum lactate value is also present in a convulsive syncope as the most important differential diagnosis to generalized epileptic seizures.

So in the present prospective study, the serum lactate concentrations are compared following convulsive and non-convulsive syncopes.

The examinations are carried out in cardiological patients who receive a tipping table examination with the aim of initiating a syncope. The question is whether there is hyperlactatemia following convulsive syncopes. If no elevated serum lactate values were measured after convulsive syncopes, this would additionally indicate the great benefit of the serum lactate value as a diagnostic marker in the generalized epileptic seizure.

In addition, a comparison is made with the parameters creatine kinase, prolactin, pH-value, bicarbonate, sodium and potassium.

If increased serum lactate values are measured following a syncope further venous blood controls are carried out at intervals of 20 minutes within the first hour and then after 90 minutes and 120 minutes until normalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with convulsive or non-convulsive syncopes
* 18 years or older

Exclusion Criteria:

* Prisoner
* Age < 18 years old
* Lack of capacity for consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cardiological patients with syncopes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the first measurements of serum lactate concentrations in blood samples between patients admitted with either a convulsive or a non-convulsive syncope | 2 hours

SECONDARY OUTCOMES:
Comparison of the first measurements of serum prolactin concentrations in blood samples between patients admitted with either a convulsive or a non-convulsive syncope | 2 hours
Comparison of the first measurements of creatine kinase concentrations in blood samples between patients with either a convulsive or a non-convulsive syncope | 2 hours
Comparison of the first measurements of pH value concentrations in blood samples between patients with either a convulsive or a non-convulsive syncope | 2 hours
Comparison of the first measurements of bicarbonate concentrations in blood samples between patients with either a convulsive or a non-convulsive syncope | 2 hours
Comparison of the first measurements of sodium and potassium concentrations in blood samples between patients with either a convulsive or a non-convulsive syncope | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Matz, Dr., Study Director — RWTH Aachen University Hospital
Locations (1):
- Department of Neurology/Department of Cardiology, University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matz O, Zdebik C, Zechbauer S, Bundgens L, Litmathe J, Willmes K, Schulz JB, Dafotakis M. Lactate as a diagnostic marker in transient loss of consciousness. Seizure. 2016 Aug;40:71-5. doi: 10.1016/j.seizure.2016.06.014. Epub 2016 Jun 23. PMID 27367837